CLINICAL TRIAL: NCT00208403
Title: Randomised, Prospective, RSA, PMS Study Comparing Acryloc™ & Palacos R in Primary Total Hip Arthroplasty
Brief Title: A Randomised Single Centre Study to Compare the Long-term Performance of Acryloc™ and Palacos® R Bone Cements in Primary Total Hip Replacement
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT02/08
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Osteoarthritis; Post-traumatic Arthritis; Avascular Necrosis
Keywords: Hip; Cement
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Acryloc™ GHV
  Interventions: Device: Acryloc™ GHV
- 2 (Active Comparator): Palacos R
  Interventions: Device: Palacos R

INTERVENTIONS:
Device: Acryloc™ GHV — A high viscosity bone cement for use in total hip replacement
  Arms: 1
Device: Palacos R — A high viscosity bone cement for use in total hip replacement
  Arms: 2

SUMMARY:
The purpose of this study is to monitor the stability of a total hip replacement within the thigh bone when used in artificial hip joints implanted with two different bone cements, Acryloc™ and Palacos® R, in the treatment of patients with hip joint disease requiring a total hip replacement. Patients who enter the study will be randomly allocated to Acryloc™ or Palacos® R and will be evaluated at regular intervals following hip surgery using patient, clinical, x-ray assessments and special x-rays which allow the stability of the hip implant to be determined

ELIGIBILITY:
Inclusion Criteria:

i) Male or female subjects, aged 60 to 75 years (inclusive), and with a weight of less than 100kg.

ii) Subjects who are able to give voluntary, written informed consent to participate in this investigation and from whom consent has been obtained.

iii) Subjects who, in the opinion of the Investigator, are able to understand this investigation, co-operate with the investigational procedures and are willing to return to the hospital for all the required post-operative follow-ups.

iv) Subjects with non-inflammatory arthritis of the hip.

v) Subjects who require a primary total hip arthroplasty and are treated at the arthroplasty section of the orthopaedics department at the Investigational Centre.

vi) Subjects who are considered suitable for a cemented femoral stem and cemented acetabular component.

Exclusion Criteria:

i) Subjects who, in the opinion of the Investigator, have an existing condition such as malignancy, severe osteoporosis, disabling musculo-skeletal problems (other than in the hips) or any other condition that would compromise their participation and follow-up in this study.

ii) Women who are pregnant.

iii) Subjects who are known drug or alcohol abusers or with psychological disorders that could effect follow-up care or treatment outcomes.

iv) Subjects who have participated in a clinical study with an investigational product in the last 6 month(s).

v) Subjects who are currently involved in any injury litigation claims.

vi) Subjects undergoing corticosteroid treatment.

vii) Subjects with any condition for whom the use of conventional bone cement is contra-indicated.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2002-10; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Distal migration of the femoral prosthesis from the time of implantation to the 2 year follow-up assessment | 2 Year

SECONDARY OUTCOMES:
Annual posterior (AP) and medio-lateral (ML) RSA translations | Annually
Merle D'Aubigne score | Annually
Radiographic analysis | Annually
Kaplan-Meier Survivorship - Revision of any component for any reason | Throughout Study

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Trondheim, Trondheim, Sor-Trondelag, Norway